CLINICAL TRIAL: NCT02871011
Title: A Blinded Placebo Controlled Clinical Trial To Evaluate Fungicidal Activity With The Topical Application Of Nitric Oxide Releasing Solution (Nors) In Subjects With Moderate To Severe Tinea Pedis (Athlete's Foot)
Brief Title: Nitric Oxide Releasing Solution (NORS) Footbath to Treat Athlete's Foot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nitric Solutions Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAN-CPT-01
Record Dates: First submitted 2016-08-04; First posted 2016-08-18 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Tinea Pedis
Keywords: Tinea Bronchodilator Agents; Tinea Pedis; Nitric Oxide; Dermatomycoses; Endothelium-Dependent Relaxing Factors; Infectious; Infection; Mycoses; Skin Diseases; Foot Dermatoses; Foot Diseases; Pruritus; Skin Manifestations Signs and Symptoms
MeSH Terms: conditions — Tinea Pedis; Dermatomycoses; Communicable Diseases; Infections; Mycoses; Skin Diseases; Foot Dermatoses; Foot Diseases; Pruritus | interventions — Nitric Oxide; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Water, delivered as a footbath for 30 minutes, daily for 3 consecutive days.
  Interventions: Drug: Water
- Nitric oxide (Experimental): Nitric oxide delivered as a footbath for 30 minutes, daily for 3 consecutive days.
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Delivered as a footbath
  Other Names: NORS
  Arms: Nitric oxide
Drug: Water — Delivered as a footbath
  Other Names: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to determine the fungicidal efficacy of nitric oxide releasing solution footbath and it's effect on the clinical signs and symptoms associated with Tinea Pedis

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Sequential Assignment Masking: Double Blind (Subject & Assessor) Primary Purpose: Treatment

ELIGIBILITY:
Inclusion Criteria:

* Positive clinical findings for moccasin, interdigital or bullous tinea pedis as determined by direct clinical examination
* Must have a clinical symptom severity score of at least 20 on a possible 64 point scale
* Written informed consent must be obtained from the subject.
* Must ≥ 19 years of age, for study sites located in British Columbia. For other locations the subject must be ≥ 18 years of age, unless local laws dictate otherwise.
* Must agree to avoid professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit until the conclusion of the trial.
* Must agree to take measures to avoid pregnancy during the 31 day study period

Exclusion Criteria:

* Has a diagnosis of either psoriasis or eczema, in or immediately around the area under evaluation.
* Has a visual diagnosis, by the investigator, of onychomycosis at a level, which in the opinion of the investigator could compromise the integrity of the study.
* Use of topical antifungals e.g. (clotrimazole, ketoconazole,miconazole, oxiconazole- (Oxistat®, Glaxo Smith Kline), sulconazole, naftifine (Naftin®, Merz), terconazole, econazole nitrate (Spectazole®, Ortho-McNeil), butoconazole ,Fluconazole, ciclopirox olamine-(Loprox®), tolnaftate, haloprogin), Zeasorb, antibacterials and corticosteroids in the preceding 5 days of screening visit (Day 1) on or immediately around the area under evaluation.
* Use of systemic corticosteroids in the preceding 7 days respectively, of screening visit (Day 1)
* Use of systemic antifungals in the preceding 7 days of screening visit (Day1) including - (terbinafine - (Lamisil®, Novartis), Itraconazole - (Sporanox®, Janssen), fluconazole- (Diflucan®, Pfizer), ketoconazole, miconazole, griseofulvin (GrisPEG®), butoconazole, terconazole, Potassium iodide)
* Has used any investigational drug(s) within 30 days preceding screening visit (Day 1)
* Is pregnant or is a nursing mother
* Is a woman of child bearing potential who is not using an adequate form of contraception (or abstinence)
* Is < 19 years of age, for study sites located in British Columbia. For other locations subject is < 18 years of age, unless local laws dictate otherwise.
* Suffers from a condition, which, in the opinion of the medical investigator, would compromise his/her safety and / or the quality of the data. Such conditions may include collagen vascular disease, diabetes mellitus, Cushing's Disease, hematological malignancy, chronic mucocutaneous candidiasis or atopy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-13 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Miller, M.D., Principal Investigator — Nitric Solutions Inc.
Locations (1):
- Fairmont Medical Clinic, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Nitric Oxide
Started | 7 | 13
Completed | 7 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Nitric Oxide | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Continuous [Mean (Full Range); unit: years] — Population: Randomized Treatment to Control of 2:1
  years | 53.1 [35 to 79] | 53.2 [34 to 79] | 53.2 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Cure: Post Treatment (Day 17)
Description: Complete cure will be determined by negative fungal culture or negative microscopic evaluation via KOH preparation and a Clinical Symptom Severity Score of ≤ 8 (0-64) on Day 17. Improvement is expressed as a lower score.
Time Frame: Day 17
Population: Intent to treat enrollment was 20 individuals but per protocol only a total of 12 participants met the criteria for both a positive fungal culture and microscopic evaluation at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Nitric Oxide
Number analyzed (Participants) | 4 | 8
Participants | 0 | 4

2. Primary Outcome: Number of Participants With Complete Cure: Post Treatment (Day 31)
Description: Complete cure will be determined by a minimum of a 12- point reduction on day 17 in the Clinical Symptom Severity Score (from >20 to <8) on a scale of 0-64. Improvement is expressed as a lower score.
Time Frame: Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Nitric Oxide
Number analyzed (Participants) | 4 | 8
Participants | 0 | 5

3. Primary Outcome: Number of Participants With Therapeutic Failure: Post Treatment (Day 17)
Description: Positive fungi colonization via mycological culture OR microscopic evaluation (KOH) AND a post treatment Clinical Symptom Severity Score of ≤ 8 (0-64) on Day 17. Improvement is expressed as a lower score.
Time Frame: Day 17
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Nitric Oxide
Number analyzed (Participants) | 4 | 8
Participants | 2 | 0

4. Primary Outcome: Number of Participants withTherapeutic Failure: Post Treatment Day 31 AND a Post Treatment Clinical Symptom Severity Score (Day 31) of < 8.
Description: Positive fungi colonization via mycological culture OR microscopic evaluation (KOH) AND a post treatment Clinical Symptom Severity Score of ≤ 8 (0-64) on Day 31. Improvement is expressed as a lower score.
Time Frame: Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Nitric Oxide
Number analyzed (Participants) | 4 | 8
Participants | 1 | 0

5. Primary Outcome: Incidence of Adverse Events
Description: Number of moderate A/E possibly related to treatment
Time Frame: Duration of the study, 31 days for each participant.
Population: Intent to treat enrollment was 20 individuals.
Measure: Number; unit: Events
Arm/Group | Control | Nitric Oxide
Number analyzed (Participants) | 7 | 13
Events | 0 | 3

6. Secondary Outcome: Change in Participants Clinical Symptom Severity Score Between Day 1 and Day 31
Description: Clinical Symptom Severity Score change in score on Day and Day 31 between all participants with an initial Clinical Symptom severity Score of >20 (0-64 scale) in the two study groups.
  Increased improvement is expressed as largest negative change and a lower score.
Time Frame: Day 1 and 31
Population: Intent to treat enrollment was 20 individuals.
Measure: Mean (Standard Deviation); unit: Clinial symptom Severity Score
Arm/Group | Control | Nitric Oxide
Number analyzed (Participants) | 7 | 13
Clinial symptom Severity Score | -3.4 (8.6) | -18.8 (7.1)

ADVERSE EVENTS:
Time Frame: Thirty-one Days
Arm/Group | Control | Nitric Oxide
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 0/7 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=7) | Nitric Oxide (N=13)
Discomfort -warm/sting (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No